CLINICAL TRIAL: NCT03142035
Title: Dienogest Versus Gonadotropin Releasing Hormone Agonist Pre-treatment in Women With Endometriosis Undergoing in Vitro Fertilization
Brief Title: Dienogest Versus GnRH-a Pre-treatment in Women With Endometriosis Undergoing IVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dina Chamsy, Assistant Professor,Minimally Invasive Gynecologic Surgery, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OGY.DC.03
Record Dates: First submitted 2017-02-22; First posted 2017-05-05 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — dienogest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dienogest (Experimental): patients will receive daily dienogest (2mg) for a total of 3 months (84 days)
  Interventions: Drug: Dienogest 2 MG; Procedure: IVF/IVF+ART
- GnRH agonist (Active Comparator): patients will receive a single GnRH-a injection (3.25mg) every 28 days for three months.
  Interventions: Drug: gonapeptyl; Procedure: IVF/IVF+ART
- Control Group (Other): patients will not receive any medical intervention and will proceed with their IFV/ICSI cycles.
  Interventions: Procedure: IVF/IVF+ART

INTERVENTIONS:
Drug: Dienogest 2 MG — Dienogest is a fourth-generation progestin of 19-nortestosterone derivative, that has been shown to improve endometriosis associated pelvic pain. It is well tolerated with no androgenic, glucocorticoid or mineralocorticoid activity. Dienogest creates a hyperprogestogenic and hypoestrogenic environment that initially induces a secretory state and then a decidualization of the ectopic endometrium and finally its atrophy. It also inhibits aromatase and COX-2 expression as well as prostaglandin E2 production in endometriotic stromal cells. It also normalizes the activity of natural killer cells and decreases the release of interleukin-1b by macrophages. These anti-inflammatory properties further help in reducing the size of endometriotic lesions
  Arms: Dienogest
Drug: gonapeptyl — gonadotropic releasing hormone agonist
  Arms: GnRH agonist
Procedure: IVF/IVF+ART — In-vitro fertilization +/- assisted reproductive technology

SUMMARY:
Endometriosis is a chronic gynecologic disease that affects approximately 10% of women in the reproductive age group . It is characterized by the presence of endometrial tissue outside the uterus, causing pelvic pain and subfertility. It is estimated that around 40% of infertile women have the diagnosis of endometriosis . Infertility secondary to endometriosis is thought to be multifactorial. Women with endometriosis often require in vitro fertilization (IVF). One medical intervention that has been shown to improve IVF outcomes in women with endometriosis is hormonal suppression with gonadotropic releasing hormone agonist (GnRH-a) for a period of 3 to 6 months .

In recent years, the effectiveness of dienogest, a fourth-generation progestin, for endometriosis treatment has been demonstrated. Dienogest seems to be as effective as GnRH-a in improving endometriosis-related pelvic pain [4]. However, no study has yet assessed whether dienogest has any benefit in treating endometriosis associated infertility.

The aim of our study is to evaluate the efficacy of dienogest versus GnRH-a in improving ongoing pregnancy rates in women undergoing IVF due to endometriosis. We will conduct a non-blinded randomized controlled trial. One group will receive dienogest 2mg daily for a period of 3 months followed by a standard IVF/Intracytoplasmic Sperm Injection (ICSI) cycle. The second group will receive one injection of 3.75mg of GnRH-a every 28 days for three doses followed by a standard IVF/ICSI cycle 3 months later. The third group will not receive any medical interventions before the planned IVF/ICSI cycle. We hypothesize that patients receiving dienogest will have similar ongoing pregnancy rates compared to patients receiving the GnRH-a injection. Secondary outcomes including number of gonadotropins consumed, number of stimulation days, number of metaphase II eggs retrieved, fertilization rate, embryo quality, miscarriage rate, clinical pregnancy rates, live birth rates and potential maternal and obstetrical complications will also be evaluated. We will also compare ongoing pregnancy rates between the groups receiving Dienogest and placebo, and GnRH agonist and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary infertility
* Endometriosis, stage III - IV, confirmed surgically by laparoscopy or laparotomy and/or radiologically by the presence of endometrioma on pelvic ultrasound or magnetic resonance imaging (MRI)
* Normal uterine cavity assessed by hysteroscopy or hysterosalpingogram
* Normal hormonal profile: TSH, prolactin, fasting blood sugar
* Normal semen analysis and mild/moderate male factor (Total motile sperm count > 5 million/ml and/or normal WHO morphology >20%)
* First IVF cycle or history of failed IVF cycles
* Washout period of ≥6 months after any diagnostic or therapeutic surgery for endometriosis or after any medical treatment with Dienogest or GnRH agonist.

Exclusion Criteria:

* • Low ovarian reserve defined by one of the following: low AMH ≤1.5ng/mL and/or basal day 3 FSH ≥ 10mIU/mL and/or basal day 3 Estradiol ≥ 60ng/mL and/or previous egg collection yield of ≤3 oocytes.

  • Absolute contraindications to dienogest, including:
* undiagnosed abnormal vaginal bleeding
* pregnancy and/or lactation
* active venous thromboembolic disorder
* history of or current arterial and cardiovascular disease (eg, MI, CVA)
* diabetes mellitus with vascular involvement
* history of or current severe hepatic disease where liver function tests remain abnormal
* history of or current hepatic neoplasia (benign or malignant)
* known or suspected sex-hormone-dependent malignancy
* ocular lesions due to ophthalmic vascular disease, such as partial or complete vision loss or defect in visual fields
* current or history of migraine with focal aura
* hypersensitivity or poor tolerance to dienogest

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 189 (Estimated)
Dates: Start 2017-10-22 (Actual); Primary Completion 2023-02-22 (Estimated); Study Completion 2023-02-22 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks of gestation
  pregnancy positive fetal cardiac activity with beyond 12 weeks of gestation (%)

SECONDARY OUTCOMES:
Gonadotropin consumption (IU) | 3 months
  Gonadotropin consumption (IU)
stimulation (days) | up to 15 days
  Duration of stimulation (days)
metaphase II oocytes retrieved | 12 weeks of gestation
  Number of metaphase II oocytes retrieved at the time of egg collection (n).
Fertilization rate | day 2
  the number of 2PN zygotes divided by the total number of mature metaphase II oocytes retrieved (%).
Embryo quality. | day 3 or 5
  Embryo quality according to embryo grading at day 3 or day5
Clinical pregnancy rate | 12 weeks of gestation
  the presence of a gestational sac, with or without cardiac activity, on ultrasound assessment (%).
Ongoing pregnancy rate -2 | 12 weeks of gestation
  pregnancy positive fetal cardiac activity with beyond 12 weeks of gestation (%)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Chamsi, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giudice LC, Kao LC. Endometriosis. Lancet. 2004 Nov 13-19;364(9447):1789-99. doi: 10.1016/S0140-6736(04)17403-5. PMID 15541453
- [Background] Strathy JH, Molgaard CA, Coulam CB, Melton LJ 3rd. Endometriosis and infertility: a laparoscopic study of endometriosis among fertile and infertile women. Fertil Steril. 1982 Dec;38(6):667-72. doi: 10.1016/s0015-0282(16)46691-4. PMID 6216124
- [Background] Sallam HN, Garcia-Velasco JA, Dias S, Arici A. Long-term pituitary down-regulation before in vitro fertilization (IVF) for women with endometriosis. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD004635. doi: 10.1002/14651858.CD004635.pub2. PMID 16437491
- [Background] Strowitzki T, Marr J, Gerlinger C, Faustmann T, Seitz C. Dienogest is as effective as leuprolide acetate in treating the painful symptoms of endometriosis: a 24-week, randomized, multicentre, open-label trial. Hum Reprod. 2010 Mar;25(3):633-41. doi: 10.1093/humrep/dep469. Epub 2010 Jan 19. PMID 20089522
- [Background] Barnhart K, Dunsmoor-Su R, Coutifaris C. Effect of endometriosis on in vitro fertilization. Fertil Steril. 2002 Jun;77(6):1148-55. doi: 10.1016/s0015-0282(02)03112-6. PMID 12057720
- [Background] Matson PL, Yovich JL. The treatment of infertility associated with endometriosis by in vitro fertilization. Fertil Steril. 1986 Sep;46(3):432-4. doi: 10.1016/s0015-0282(16)49581-6. PMID 3091408
- [Background] Simon C, Gutierrez A, Vidal A, de los Santos MJ, Tarin JJ, Remohi J, Pellicer A. Outcome of patients with endometriosis in assisted reproduction: results from in-vitro fertilization and oocyte donation. Hum Reprod. 1994 Apr;9(4):725-9. doi: 10.1093/oxfordjournals.humrep.a138578. PMID 8046030
- [Background] Cahill DJ, Wardle PG, Maile LA, Harlow CR, Hull MG. Ovarian dysfunction in endometriosis-associated and unexplained infertility. J Assist Reprod Genet. 1997 Nov;14(10):554-7. doi: 10.1023/a:1022568331845. PMID 9447453
- [Background] Norenstedt SN, Linderoth-Nagy C, Bergendal A, Sjoblom P, Bergqvist A. Reduced developmental potential in oocytes from women with endometriosis. J Assist Reprod Genet. 2001 Dec;18(12):644-9. doi: 10.1023/a:1013111200251. PMID 11808845
- [Background] Nakahara K, Saito H, Saito T, Ito M, Ohta N, Takahashi T, Hiroi M. Ovarian fecundity in patients with endometriosis can be estimated by the incidence of apoptotic bodies. Fertil Steril. 1998 May;69(5):931-5. doi: 10.1016/s0015-0282(98)00038-7. PMID 9591505
- [Background] Pellicer A, Albert C, Mercader A, Bonilla-Musoles F, Remohi J, Simon C. The follicular and endocrine environment in women with endometriosis: local and systemic cytokine production. Fertil Steril. 1998 Sep;70(3):425-31. doi: 10.1016/s0015-0282(98)00204-0. PMID 9757870
- [Background] Toya M, Saito H, Ohta N, Saito T, Kaneko T, Hiroi M. Moderate and severe endometriosis is associated with alterations in the cell cycle of granulosa cells in patients undergoing in vitro fertilization and embryo transfer. Fertil Steril. 2000 Feb;73(2):344-50. doi: 10.1016/s0015-0282(99)00507-5. PMID 10685541
- [Background] Garcia-Velasco JA, Mulayim N, Kayisli UA, Arici A. Elevated soluble Fas ligand levels may suggest a role for apoptosis in women with endometriosis. Fertil Steril. 2002 Oct;78(4):855-9. doi: 10.1016/s0015-0282(02)03320-4. PMID 12372468
- [Background] Vercellini P, Somigliana E, Vigano P, Abbiati A, Barbara G, Crosignani PG. Surgery for endometriosis-associated infertility: a pragmatic approach. Hum Reprod. 2009 Feb;24(2):254-69. doi: 10.1093/humrep/den379. Epub 2008 Oct 23. PMID 18948311
- [Background] Geber S, Ferreira DP, Spyer Prates LF, Sales L, Sampaio M. Effects of previous ovarian surgery for endometriosis on the outcome of assisted reproduction treatment. Reprod Biomed Online. 2002 Sep-Oct;5(2):162-6. doi: 10.1016/s1472-6483(10)61619-7. PMID 12419041
- [Background] Aboulghar MA, Mansour RT, Serour GI, Al-Inany HG, Aboulghar MM. The outcome of in vitro fertilization in advanced endometriosis with previous surgery: a case-controlled study. Am J Obstet Gynecol. 2003 Feb;188(2):371-5. doi: 10.1067/mob.2003.13. PMID 12592242
- [Background] Tei C, Miyazaki T, Kuji N, Tanaka M, Sueoka K, Yoshimura Y. Effect of danazol on the pregnancy rate in patients with unsuccessful in vitro fertilization-embryo transfer. J Reprod Med. 1998 Jun;43(6):541-6. PMID 9653702
- [Background] Marcus SF, Edwards RG. High rates of pregnancy after long-term down-regulation of women with severe endometriosis. Am J Obstet Gynecol. 1994 Sep;171(3):812-7. doi: 10.1016/0002-9378(94)90103-1. PMID 8092234
- [Background] Chedid S, Camus M, Smitz J, Van Steirteghem AC, Devroey P. Comparison among different ovarian stimulation regimens for assisted procreation procedures in patients with endometriosis. Hum Reprod. 1995 Sep;10(9):2406-11. doi: 10.1093/oxfordjournals.humrep.a136308. PMID 8530675
- [Background] Ruiz-Velasco V, Allende S. Goserelin followed by assisted reproduction: results in infertile women with endometriosis. Int J Fertil Womens Med. 1998 Jan-Feb;43(1):18-23. PMID 9532465
- [Background] Bizzarri N, Remorgida V, Leone Roberti Maggiore U, Scala C, Tafi E, Ghirardi V, Salvatore S, Candiani M, Venturini PL, Ferrero S. Dienogest in the treatment of endometriosis. Expert Opin Pharmacother. 2014 Sep;15(13):1889-902. doi: 10.1517/14656566.2014.943734. Epub 2014 Jul 29. PMID 25069386
- [Background] Klipping C, Duijkers I, Remmers A, Faustmann T, Zurth C, Klein S, Schuett B. Ovulation-inhibiting effects of dienogest in a randomized, dose-controlled pharmacodynamic trial of healthy women. J Clin Pharmacol. 2012 Nov;52(11):1704-13. doi: 10.1177/0091270011423664. Epub 2011 Nov 29. PMID 22128200
- [Background] Surrey ES, Silverberg KM, Surrey MW, Schoolcraft WB. Effect of prolonged gonadotropin-releasing hormone agonist therapy on the outcome of in vitro fertilization-embryo transfer in patients with endometriosis. Fertil Steril. 2002 Oct;78(4):699-704. doi: 10.1016/s0015-0282(02)03373-3. PMID 12372443